CLINICAL TRIAL: NCT01625507
Title: The Alberta Diet: a Proposal for Its Implementation
Brief Title: The Alberta Diet: Effectiveness Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RES0013109
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PANDA intervention (Experimental): 12 week nutritional intervention, including 6 classroom/community sessions, plus two sample collection visits.
  Interventions: Behavioral: PANDA intervention

INTERVENTIONS:
Behavioral: PANDA intervention — Participants will follow a menu plan and receive training in how to manage their diet in type 2 diabetes, following the recommendations of the Canadian Diabetes Association, 2008

SUMMARY:
The study hypothesis is that individuals with type 2 diabetes (T2D), who adhere to the PANDA intervention, will have improved compliance with the nutritional therapy recommendations of the Canadian Diabetes Association. Specific objectives of this proposal: The objectives of the investigators PANDA (Physical Activity and Nutrition for Diabetes in Alberta) are to (a) to devise and evaluate the efficacy of a multi-level, practical, nutrition intervention program that promotes the individual factors required for effective self-management practices AND that explicitly incorporate strategies to improve food availability, accessibility and acceptability and (b) to use these interventions as a means to examine the relationships between food availability, accessibility, acceptability, adherence to Nutrition Therapy Guidelines, and metabolic indicators of diabetes control in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, and speak/write English.
* Have attended a diabetes education session delivered by their healthcare provider.

Exclusion Criteria:

* Participants with type 1 diabetes, and those who are unable to speak English.
* People with end-stage renal disease or gastrointestinal diseases that require specialized diets will also be excluded.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine B Chan, PhD, Principal Investigator — University of Alberta
Locations (1):
- Alberta Diabetes Institute, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- PANDA Intervention: 12 week nutritional intervention, including 6 classroom/community sessions, plus two sample collection visits.
  PANDA intervention: Participants will follow a menu plan and receive training in how to manage their diet in type 2 diabetes (T2D), following the recommendations of the Canadian Diabetes Association, 2008
Period: Overall Study
Arm/Group | PANDA Intervention
Started | 73
Completed | 63
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | PANDA Intervention
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.7)
Gender [Count of Participants; unit: Participants]
  Female | 34
  Male | 39
Region of Enrollment [Number; unit: participants]
  Canada | 73
Education [Number; unit: participants]
  Less than high school | 5
  High school completed | 28
  College or university degree | 40
Employment [Number; unit: participants]
  Wages and salaries | 41
  Self-employment | 5
  Retired | 18
  Unemployed | 2
  Other | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Energy Intake
Description: Measured using repeated 24 hour dietary recalls (pre and post-intervention)
Time Frame: 4 months
Population: All participants, intention to treat protocol
Measure: Mean (95% Confidence Interval); unit: kcal
Groups:
- All Participants: T2D patients comparing post- to pre-intervention
Arm/Group | All Participants
Number analyzed (Participants) | 73
kcal | -178 [-305 to -51]

2. Primary Outcome: Change in Macronutrient Intake
Description: Measured using repeated 24 hour dietary recalls (pre and post-intervention)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: percentage of total energy
Arm/Group | All Participants
Number analyzed (Participants) | 73
percentage of total energy
  Total fat | -1 [-3 to 0]
  Saturated fat | 0 [-1 to 0]
  Protein | 0 [0 to 1]
  Carbohydrate | 2 [0 to 4]
  Added sugar | 0 [-1 to 1]

3. Primary Outcome: Change in Nutrient Intake
Description: Measured using repeated 24 hour dietary recalls (pre and post-intervention)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: grams
Arm/Group | All Participants
Number analyzed (Participants) | 73
grams
  Total fat | -10 [-18 to -3]
  Saturated fat | -3 [-6 to -1]
  Monounsaturated fat | -3 [-6 to 0]
  Polyunsaturated fat | 0 [-2 to 2]
  Protein | -6 [-11 to 0]
  Carbohydrate | -12 [-28 to 4]
  Fiber | 0 [-1 to 1]
  Total sugar | -5 [-13 to 2]
  Added sugar | -9 [-17 to 0]
  Cholesterol | -.003 [-.045 to .05]
  Sodium | -.572 [-.869 to -.275]

4. Secondary Outcome: Change in Hemoglobin A1c
Description: a surrogate of blood glucose control
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: percentage of hemoglobin A1c
Arm/Group | All Participants
Number analyzed (Participants) | 73
percentage of hemoglobin A1c | -0.7 [-1 to -0.4]

5. Secondary Outcome: Program Retention
Description: attendance at meetings
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | PANDA Intervention
Number analyzed (Participants) | 73
Participants | 63

6. Secondary Outcome: Change in Body Mass Index
Description: Actual weight and height used to calculate BMI pre- and post-intervention
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: kg/m2
Arm/Group | All Participants
Number analyzed (Participants) | 73
kg/m2 | -0.6 [-0.8 to -0.4]

7. Secondary Outcome: Body Composition
Description: body fat and fat-free mass
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | All Participants
Number analyzed (Participants) | 73
percentage change from baseline
  Change in Fat mass % | -0.8 [-1.5 to 0]
  Change in Fat free mass % | 0.8 [0.1 to 1.6]

8. Secondary Outcome: Change in Blood Biomarkers
Description: blood lipids: triglyceride, total cholesterol, LDL-cholesterol, HDL-cholesterol
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 73
mg/dL
  Total cholesterol | -63.5 [-80.1 to -46.9]
  High density lipoprotein cholesterol | 27.5 [20.2 to 34.8]
  Low density lipoprotein cholesterol | -88.9 [-105.3 to -72.5]
  Triglycerides | -10.4 [-23.1 to 2.2]

9. Secondary Outcome: Change in Perceived Dietary Adherence Questionnaire Score
Description: Questionnaire assessing self-reported adherence to 9 criteria, whose individual scores (range 0-7) are summed to get the total score. Maximum total score is 63. Minimum total score is 0. A higher score means higher dietary adherence.
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 73
units on a scale | 9.3 [5.4 to 12.9]

10. Secondary Outcome: Food Acceptability
Description: questionnaire based on items related to personal and cultural acceptability of the recommended diet
Time Frame: 4 months
Reporting Status: Not Posted

11. Secondary Outcome: Food Accessibility
Description: questionnaire of items related to financial and physical accessibility of foods in the diet recommended for diabetes
Time Frame: 4 months
Reporting Status: Not Posted

12. Secondary Outcome: Food Availability
Description: questionnaire of items related to the availability in local stores of the food items recommended in the diet for diabetes.
Time Frame: 4 months
Reporting Status: Not Posted

13. Secondary Outcome: Change in Waist Circumference
Description: Measured using repeated 24 hour dietary recalls (pre and post-intervention
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 73
cm | -2.4 [-3.0 to -1.8]

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Groups:
- All Participants: T2D diabetes patients
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No